CLINICAL TRIAL: NCT07241195
Title: Study on the Construction of Disease Cohort for Fatty Liver in the Elderly and Its Prevention and Treatment Strategies
Brief Title: A Community-based Prospective Cohort Study on Metabolic Dysfunction-Associated Fatty Liver Disease in Older Adults: From Metabolic Trajectories to Extrahepatic Outcomes
Acronym: MAPS Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: SJP20250401
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: NAFLD and NASH; NAFLD( Non-alcoholic Fatty Liver Disease ); NAFLD Cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group
- Observation Group: Lifestyle interventions

SUMMARY:
To establish a cohort of elderly fatty liver disease based on the community medical examination population. Through the large-scale cohort study, the risk factors affecting fatty liver in the elderly will be explored in depth from the aspects of lifestyle, environment and genetics, the development pattern and mechanism of fatty liver in the elderly will be analysed, and the health risk assessment system and Chinese standard for fatty liver in the elderly covering cardiovascular risk, risk of hepatic fibrosis and risk of sarcopenia will be established, so as to provide the scientific basis for the precise intervention of fatty liver in the elderly in China.

ELIGIBILITY:
Inclusion Criteria:

* ① Elderly people aged ≥65 years among permanent residents (living for more than 5 years) in the survey area;

  * Imaging diagnosis (ultrasound or FibroScan/FibroTouch) of fatty liver; -③ Voluntary participation in this study and signing an informed consent form.

Exclusion Criteria:

* ①Major disability, mental illness, major wasting disease, severe cardiac, pulmonary and renal insufficiency;

  * Patients with combined primary liver cancer or other types of cancer; -③Patients who have received liver transplant or other organ transplants.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: elder people
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2026-03-12 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of liver fibrosis | 2 years

SECONDARY OUTCOMES:
Incidence of cardiovascular disease | 2 years
Incidence of sarcopenia | 2 years

IPD SHARING:
Plan to Share IPD: No